CLINICAL TRIAL: NCT06567327
Title: A Two-Part Phase 1, Open-Label, Fixed-Sequence Study to Evaluate the Multiple Dose Pharmacokinetics of Danuglipron Following Oral Administration and The Effects of Steady-State Danuglipron on the Pharmacokinetics of Single Oral Dose of Atorvastatin and Rosuvastatin in Otherwise Healthy Adult Participants With Overweight or Obesity
Brief Title: A Study to Learn How the Study Medicine Danuglipron is Taken Up Into the Blood and If Danuglipron Changes How the Body Processes Other Study Medicines (Atorvastatin and Rosuvastatin) in Healthy Adults Who Are Overweight or Obese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C3421086; NCT06567327 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-08-09; First posted 2024-08-22 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Obesity
Keywords: Overweight; Obesity; Danuglipron; GLP-1; Drug-drug interaction; Overtly healthy; Atorvastatin; Rosuvastatin
MeSH Terms: conditions — Obesity; Overweight | interventions — danuglipron; Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Participants will receive a single dose of atorvastatin and multiple oral doses of danuglipron with and without atorvastatin
  Interventions: Drug: Danuglipron; Drug: Atorvastatin
- Cohort 2 (Experimental): Participants will receive a single dose of rosuvastatin and multiple oral doses of danuglipron with and without rosuvastatin
  Interventions: Drug: Danuglipron; Drug: Rosuvastatin
- Cohort 3 (Experimental): Participants will receive a single dose of atorvastatin and multiple oral doses of danuglipron with and without atorvastatin
  Interventions: Drug: Danuglipron; Drug: Atorvastatin
- Cohort 4 (Experimental): Participants will receive a single dose of rosuvastatin and multiple oral doses of danuglipron with and without rosuvastatin
  Interventions: Drug: Danuglipron; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Danuglipron — Danuglipron oral tablets
  Other Names: PF-06882961
Drug: Atorvastatin — Atorvastatin oral tablets
  Arms: Cohort 1; Cohort 3
Drug: Rosuvastatin — Rosuvastatin oral tablets
  Arms: Cohort 2; Cohort 4

SUMMARY:
The purpose of this study is to learn the following about the study medicine, danuglipron, after multiple days of dosing in healthy adults who are overweight or obese:

* how the study medicine, danuglipron, is taken up into the blood
* if the study medicine, danuglipron, changes how the body processes other study medicines (Atorvastatin and Rosuvastatin)
* about the safety and tolerability of danuglipron

The study will take place in 4 Cohorts (groups). The total number of weeks of the study is about 23 (about 6 months) for Cohort 1 and 22 weeks (about 5.5 months) for Cohort 2, 21 weeks (about 5 months) for Cohort 3 and 20 weeks (about 5 months) for Cohort 4.

ELIGIBILITY:
Key Inclusion Criteria:

* 18 to < 65 years of age
* Body mass index (BMI) of ≥25.0-45.4 kg/m2; and a total body weight >50 kg (110 lb)

Key Exclusion Criteria:

* Evidence or history of any clinically significant medical conditions or laboratory abnormality
* Any condition possibly affecting drug absorption
* Known intolerance/hypersensitivity to a GLP-1R agonist and/or known hypersensitivity or contraindication to atorvastatin (Cohort 1 and 3 participants) or rosuvastatin (Cohort 2 and 4 participants)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2024-08-28 (Actual); Primary Completion 2025-03-16 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Steady-state area under the concentration-time profile from time zero to 24 hours (AUC24) for danuglipron | Predose to 24 hours post danuglipron administration
Steady-state maximum observed concentration (Cmax) for danuglipron | Predose to 24 hours post danuglipron administration
Steady-state time to reach maximum observed concentration (Tmax) for danuglipron | Predose to 24 hours post danuglipron administration
Area under the concentration-time curve from time zero extrapolated to infinite time (AUCinf), as data permit, for atorvastatin | Predose to 72 hours post atorvastatin administration
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) for atorvastatin (only if AUCinf is not reportable) | Predose to 72 hours post atorvastatin administration
Area under the concentration-time curve from time zero extrapolated to infinite time (AUCinf), as data permit, for rosuvastatin | Predose to 96 hours post rosuvastatin administration
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) for rosuvastatin (only if AUCinf is not reportable) | Predose to 96 hours post rosuvastatin administration

SECONDARY OUTCOMES:
Number of participants reporting Treatment Emergent Adverse Events (TEAEs) | From baseline up to 28-35 days post last dose taken
Number of participants reporting clinically significant clinical laboratory abnormalities | From baseline up to 28-35 days post last dose taken
Number of participants reporting clinically significant vital sign abnormalities | From baseline up to 28-35 days post last dose taken
Change from baseline in body weight | From baseline up to 28-35 days post last dose taken
Number of participants reporting clinically significant changes ECG abnormalities | From baseline up to 28-35 days post last dose taken

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Qps - Mra, Llc., South Miami, Florida
  - Qps-Mra, Llc, South Miami, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3421086